CLINICAL TRIAL: NCT06215989
Title: Treatment of ACuTe Coronary Syndromes With Low-dose colchICine (TACTIC): a Randomised, Double-blinded, Placebo-controlled, Multicentric Trial
Brief Title: Treatment of ACuTe Coronary Syndromes With Low-dose colchICine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TACTIC
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Acute Coronary Syndrome; Unstable Angina; ST Elevation Myocardial Infarction; Non ST Segment Elevation Myocardial Infarction; Colchicine
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; ST Elevation Myocardial Infarction | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine group (Experimental): Patients are randomized within 48 hours after diagnosis of ACS, and on the day of randomization, eligible patients undergo standard treatment plus colchicine (0.5mg qd from 1st month to 12th month).
  Interventions: Drug: Colchicine Pill
- Placebo group (Placebo Comparator): Patients are randomized within 48 hours after diagnosis of ACS, and on the day of randomization, eligible patients undergo standard treatment plus placebo (1 tablet qd from 1st month to 12th month).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine Pill — Colchicine 0.5mg once daily will be given on the basis of standard treatment of ACS recommended by guidelines
  Other Names: Colchicine 0.5 MG
  Arms: Colchicine group
Drug: Placebo — Placebo one tablet once daily will be given on the basis of standard treatment of ACS recommended by guidelines
  Arms: Placebo group

SUMMARY:
This trial is designed to evaluate whether low-dose colchicine, in addition to standard treatment recommended by guidelines, further reduces the risk of major adverse cardiovascular events in patients with acute coronary syndromes (ACS) through a prospective, randomized, double-blind, placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Background: Colchicine is a cheap and potent oral anti-inflammatory drug that can exert its anti-inflammatory effect on the pathogenesis of ACS. The 2023 updated guidelines for the management of chronic stable coronary artery disease (SCAD) by the American Heart Association (AHA)/American College of Cardiology (ACC) have identified colchicine as the drug of choice for secondary preventive treatment in patients with SCAD to reduce the risk of recurrence of adverse cardiovascular events. Despite the current optimal medical therapies, some ACS patients still suffer recurrent adverse cardiovascular events and mortality. Existing clinical studies have not fully clarified whether early use of colchicine to reduce inflammatory responses is associated with greater clinical benefit after ACS. The effect of colchicine on cardiovascular outcomes in the ACS patients needs further elucidation.

Methods: Patients aged 18 years and older with a definite diagnosis of ACS are randomly assigned to two groups in a 1:1 ratio after signing the informed consent form. Colchicine group: standard treatment + colchicine (0.5mg qd) from 1st month to 12th month after randomization. Placebo group: standard treatment + placebo (1 tablet qd) from 1st month to 12th month after randomization. The primary endpoint is the composite of cardiovascular death, non-fatal ischemic stroke, non-fatal spontaneous (non-operation related) myocardial infarction, readmission for ACS, and ischaemia driven (unplanned) revascularization at 1 year after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Definite diagnosis of ACS;
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Type 2 myocardial infarction (Patients with symptoms or signs of myocardial ischemia and evidence of increased oxygen demand or decreased supply [for example, tachyarrhythmia, hypotension, or anaemia] secondary to an alternative pathology and myocardial necrosis are defined as suffering type 2 myocardial infarction. The classification of type 2 myocardial infarction also includes patients with coronary vasospasm, embolism or spontaneous dissection without evidence of atherothrombosis related to coronary artery disease);
* Valvular heart disease that is considered likely to require surgical intervention;
* History of non-skin cancer in the past 3 years;
* Inflammatory bowel disease or chronic diarrhea;
* History of gastric ulcer or previous gastric bleeding;
* Neuromuscular diseases or non-transient (At least 2 laboratory tests) creatine kinase levels greater than 3 times the upper limit of the normal range (except those associated with myocardial infarction);
* Clinically significant non-transient (At least 2 laboratory tests) blood abnormalities(Hemoglobin <100g/L or hematocrit < 30% or > 52% or white blood cell count < 3×109/L or platelet count < 100×109/L);
* Estimated glomerular filtration rate (eGFR)<30mL/min/1.73m2 (based on CKD-EPI formula);
* Serum alanine aminotransferase and/or aspartate aminotransferase levels greater than 2 times the upper limit of the normal range accompanied by serum total bilirubin levels greater than 2 times the upper limit of the normal range or severe liver disease with coagulation disorders(INR>1.5)(except for elevated glutamic oxalacetic transaminase associated with myocardial infarction);
* Decline in cognitive function due to inability to perform basic activities of daily living independently;
* Drug or alcohol abuse;
* Other immunosuppressive therapies already in existence or planned;
* Other causes require long-term colchicine treatment;
* History of clear or suspected colchicine allergy;
* Strong CYP3A4 or P-glycoprotein inhibitors (such as cyclosporine, antiretrovirals, antifungals, erythromycin and clarithromycin) have been used and no other alternative drugs can be used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6574 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 1 year after randomization
  Rate of the composite of cardiovascular death, non-fatal ischemic stroke, non-fatal spontaneous (non-operation related) myocardial infarction, readmission for ACS, and ischaemia driven (unplanned) revascularization

SECONDARY OUTCOMES:
Key secondary endpoint | 1 year after randomization
  Rate of the composite of cardiovascular death, non-fatal ischemic stroke, and non-fatal spontaneous (non-operation related) myocardial infarction
Secondary endpoint 1 | 1 year after randomization
  Rate of all-cause death
Secondary endpoint 2 | 1 year after randomization
  Rate of cardiovascular death
Secondary endpoint 3 | 1 year after randomization
  Rate of non-fatal ischemic stroke
Secondary endpoint 4 | 1 year after randomization
  Rate of non-fatal spontaneous (non-operation related) myocardial infarction
Secondary endpoint 5 | 1 year after randomization
  Readmission rate for ACS
Secondary endpoint 6 | 1 year after randomization
  Rate of ischaemia-driven (unplanned) revascularization
Secondary endpoint 7 | 1 year after randomization
  Rate of type 3-5 bleeding events as defined by the BARC bleeding criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, PhD, MD, Study Chair — Beijing Anzhen Hospital; Xiaoli Liu, PhD, MD, Study Director — Beijing Anzhen Hospital; Xiaoteng Ma, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No